CLINICAL TRIAL: NCT00098761
Title: Phase I Study Of Cloretazine (VNP40101M) In Children With Recurrent, Progressive Or Refractory Primary Brain Tumors
Brief Title: VNP40101M in Treating Young Patients With Recurrent, Progressive, or Refractory Primary Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000396779; PBTC-017; VION-VNP40101M
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood brain stem glioma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; childhood central nervous system germ cell tumor; childhood choroid plexus tumor; childhood craniopharyngioma; childhood infratentorial ependymoma; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Optic Nerve Glioma; Astrocytoma; Familial ependymoma; Medulloblastoma; Choroid Plexus Neoplasms | interventions — laromustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: laromustine — This is a dose escalation study. Participants receive 20, 30, 45, 60, 78, 103, 137, 182, or 242 mg/m2/day intravenously over 30 minutes for 5 consecutive days every 6 weeks up to 48 weeks.
  Other Names: Cloretazine; VNP40101M

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as VNP40101M, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of VNP40101M in treating young patients with recurrent, progressive, or refractory primary brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of VNP40101M in pediatric patients with recurrent, progressive, or refractory primary brain tumors.

Secondary

* Determine the pharmacokinetics of this drug and its active metabolite VNP4090CE in these patients.
* Determine the efficacy of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to receiving ≥ 1 of the following prior therapies: craniospinal irradiation (yes vs no), autologous bone marrow transplant (yes vs no), and > 2 myelosuppressive chemotherapy or myelosuppressive biologic therapy regimens (yes vs no).

Patients receive VNP40101M IV over 30 minutes on days 1-5. Treatment repeats every 42 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 2-6 patients per stratum receive escalating doses of VNP40101M until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 25% of patients experience dose-limiting toxicity. A total of 12 patients are treated at the MTD.

Patients are followed for 3 months.

PROJECTED ACCRUAL: A total of 4-60 patients (2-30 per stratum) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* primary brain tumor, including benign brain tumors (e.g., low-grade glioma)

  * Recurrent or progressive disease OR refractory to standard therapy NOTE: *Patients with intrinsic brain stem or diffuse optic pathway tumors do not require histological confirmation, but must have clinical and/or radiographic evidence of disease progression
* No bone marrow disease

PATIENT CHARACTERISTICS:

Age

* 21 and under

Performance status

* Karnofsky 50-100% (for patients > 16 years of age) OR
* Lansky 50-100% (for patients ≤ 16 years of age)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3*
* Platelet count ≥ 100,000/mm^3*
* Hemoglobin ≥ 8 g/dL* NOTE: *Unsupported

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* No overt hepatic disease

Renal

* BUN < 25 mg/dL
* Creatinine ≤ 1.5 times ULN for age OR
* Glomerular filtration rate > 70 mL/min
* No overt renal disease

Cardiovascular

* Shortening fraction ≥ 30% by echocardiogram OR
* Ejection fraction ≥ 50% by gated radionucleotide study
* No clinically significant cardiac arrhythmia by EKG
* No overt cardiac disease

Pulmonary

* DLCO ≥ 60% of predicted
* Chest X-ray normal (defined as absence of pulmonary infiltrates, pneumonitis, pleural effusion, pulmonary hemorrhage, or fibrosis) AND a resting pulse oximetry reading of > 94% in room air (for patients who cannot perform the DLCO)
* No overt pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Neurologic deficits allowed provided there has been no deficit progression for ≥ 1 week before study entry
* No uncontrolled infection
* No known hypersensitivity to polyethylene glycol

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 6 months since prior allogeneic bone marrow or stem cell transplantation
* At least 3 months since prior autologous bone marrow or stem cell transplantation
* More than 1 week since prior colony-stimulating factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or epoetin alfa)
* At least 3 weeks since prior myelosuppressive anticancer biologic therapy
* No concurrent routine colony-stimulating factors

Chemotherapy

* At least 3 weeks since prior myelosuppressive anticancer chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* Concurrent corticosteroids allowed provided dose is stable or decreasing for ≥ 1 week before study entry

Radiotherapy

* At least 3 months since prior craniospinal irradiation ≥ 18 Gy
* At least 2 weeks since prior focal irradiation to the primary tumor and/or symptomatic metastatic sites

Surgery

* Not specified

Other

* At least 7 days since prior nonmyelosuppressive anticancer therapy
* At least 7 days since prior investigational agents
* Concurrent enzyme-inducing anticonvulsant drugs allowed
* No other concurrent anticancer or experimental agents or therapies

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2005-02; Primary Completion 2006-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Estimate the maximum tolerated dose | First 6 weeks of therapy
Number of participants with dose limiting toxicities | First 6 weeks of therapy

SECONDARY OUTCOMES:
Pharmacokinetics | Day 1 of therapy
  Plasma samples for pharmacokinetic studies will be collected with the first dose of the study drug pre-infusion, and 5, 15, and 30 minutes, 1 hour, 2 hours, and 4 hours after the end of infusion. VNP40101M plasma concentration-time data will be modeled and the individual pharmacokinetic pararmeters volume of the central compartment, elimination rate constant, and half-life will be estimated.
Tumor response to VNP40101M | Prior to course 3, 5, and 7 and end of therapy
  MRI of the brain will be obtained prior to couses 3, 5, and 7 and at the end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sri Gururangan, MRCP (UK), Study Chair — Duke University
Locations (10):
- United States (10):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Gururangan S, Turner CD, Stewart CF, O'Shaughnessy M, Kocak M, Poussaint TY, Phillips PC, Goldman S, Packer R, Pollack IF, Blaney SM, Karsten V, Gerson SL, Boyett JM, Friedman HS, Kun LE. Phase I trial of VNP40101M (Cloretazine) in children with recurrent brain tumors: a pediatric brain tumor consortium study. Clin Cancer Res. 2008 Feb 15;14(4):1124-30. doi: 10.1158/1078-0432.CCR-07-4242. PMID 18281546